CLINICAL TRIAL: NCT06826404
Title: The Effects of Using High-fidelity Simulators and Standardized Patients on the Stoma Care Skills and Learning Satisfaction Level on Nursing Students: A Randomized Controlled Trial
Brief Title: High-fidelity Simulators and Standardized Patients on the Stoma Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, Research Assistant Doctor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Wearable Ostomy Model
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Simulation-based Learning; Nursing Students; Ostomy
Keywords: Nursing students; Simulation; Ostomy care

STUDY DESIGN:
Intervention Model Description: Nursing students who were to be taught stoma care skills with a standardized patient vs. low-fidelity simulator included in the study were randomly assigned to a study and a control group (1:1 randomization).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Standardized patient with weareble ostomy model) (Experimental): The study group will be taught stoma care skills with a standardized patient wearing a wearable ostomy model.
  Interventions: Device: Training provided with a wearable ostomy model and standardized patient
- Control group (Low fidelity simulator) (Active Comparator): The study group will be taught stoma care skills with a low fidelity simulator.
  Interventions: Other: Training low fidelity simulator

INTERVENTIONS:
Device: Training provided with a wearable ostomy model and standardized patient — The subjects of what is stoma, nursing care after stoma surgery, and care of the peristomal area will be explained to the students participating in the study theoretically by the responsible director in a session and for a maximum of 30 minutes with plain narration and discussion methods, not exceeding 30 slides. Both groups will receive this training at the same time. After this explanation, stoma care will be performed on a wearable colostomy model by a volunteer student who is doing her doctorate in Surgical Diseases Nursing in accordance with the skill guide "Changing the Ostomy Bag and Nursing Care of the Peristomal Area" developed by the director of the study based on literature, and nursing students will be given the opportunity to ask questions, and then the skill will be demonstrated twice on the wearable stoma model by following the steps in the learning guide.
  Arms: Intervention group (Standardized patient with weareble ostomy model)
Other: Training low fidelity simulator — The subjects of what is stoma, nursing care after stoma surgery, and care of the peristomal area will be explained to the students participating in the study theoretically by the responsible facilitator in one session and for a maximum of 30 minutes, using plain narration and discussion methods, not exceeding 30 slides. Both groups will receive this training at the same time. After this explanation, skill training will be carried out on a lifeless mannequin in accordance with the skill guide "Changing the Ostomy Bag and Nursing Care of the Peristomal Area" developed by the facilitator of the study based on literature.
  Arms: Control group (Low fidelity simulator)

SUMMARY:
This is a randomized controlled study to investigate the effects of skill training on a low-fidelity simulator with a standardized patient using a wearable ostomy model on the stoma care skills and satisfaction levels of nursing students.

DETAILED DESCRIPTION:
Phase 1: Design of wearable colostomy model The wearable colostomy model to be designed within the scope of the project will be soft, skin-sensitive, in accordance with the real anatomy and will have wearable qualities with the help of hanger-velcro tape. There will be one healthy and normal-looking stoma on the model. The velcro tape system of the model will be made of elastic and adjustable velcro tapes according to waist measurements and will be placed on the back of the belt. The width of the tape system will be 5 cm and the length will be 90 cm. The hooked part of the velcro tapes will be fixed to one end of the elastic belt and the looped part will be fixed to the other end, the looped part will be kept longer and the belt will be adjustable at different lengths. The velcro tapes will be placed on the fabric and will be joined by sewing. On this system, a soft skin-colored medical silicone human skin will be made by sewing or gluing the abdominal surface. A dark pink stoma appearance will be created on this abdominal surface, with a diameter of 2.5 cm, slightly raised and natural from the skin surface. Modeling clay will be used to create this appearance.

Phase 2: Wearable colostomy model stoma care training What is a stoma, nursing care after stoma surgery, peristomal area care will be explained to the students participating in the study theoretically by the responsible facilitator in one session and for a maximum of 30 minutes with plain narration and discussion methods, not exceeding 30 slides. Both groups will receive this training at the same time. After this explanation, the skill guide "Changing the Ostomy Bag and Nursing Care of the Peristomal Area" developed by the facilitator of the study based on literature will be developed. This guide will be sent to 5 academicians who are experts in the field of Surgical Disease Nursing, expert opinions will be received and the skill learning guide will be finalized in line with the opinions received. According to the skill steps in this learning guide, the researcher will perform stoma care on a wearable colostomy model by a volunteer student who is doing her doctorate in Surgical Diseases Nursing and will provide nursing students with the opportunity to ask questions, then she will be provided with the opportunity to demonstrate the skill on the wearable stoma model twice by following the steps in the learning guide. The same process will be performed with the other group on an inanimate mannequin and with the same steps. In the study, one group will perform the skill with a wearable ostomy model, while the other group will teach the skill on an inanimate mannequin with an ostomy. Skill teaching will be planned on different days and times, and the level of interaction between the groups regarding the skill teaching will be minimized.

Phase 3: Evaluation of nursing students' stoma care skills, satisfaction with the simulation experience and their recommendations All students will perform the skill on a standard patient with a wearable ostomy model. This process will be conducted by an independent researcher. This scoring and evaluation will take place in a laboratory environment. After scoring, the simulation experience satisfaction scale will be given to the students and they will be asked to fill it out.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completing the Internal Medicine Nursing course
* Taking the Surgical Disease Nursing course
* Not having any absences from the 7th week (the week when the
* Gastrointestinal System Surgery topic is covered)
* Participating in the study process completely

Exclusion Criteria:

* Retaking Surgical Nursing course due to failure
* Participating in a different skill course related to stoma care
* Having provided stoma care at any time before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Stoma care skill points | Within 3 weeks after stoma care skill teaching
  The key developed by İncesu and his colleagues consists of 23 items. The items in the key include the gradual steps of stoma care such as explaining the procedure to the patient, preparing the materials, and protecting privacy regarding the students' stoma care skills. The key is planned as 'insufficient' (0 points) if the practitioner cannot perform the application by observing the student or does it wrong, 'partially sufficient' (1 point) if the step is applied correctly but in the wrong order, and 'sufficient' (2 points) if the step is applied correctly and in the wrong order. The minimum score to be obtained from the key is 0, and the maximum score is 46. Although there is no cut-off value for the scale, it is interpreted that the care skill increases as the score obtained increases. The scale will be applied once by an independent evaluator after the skill training for all students.
Simulation experience satisfaction level | Within 3 weeks after stoma care skill teaching
  The scale developed by Tüzer and his colleagues consists of three sub-dimensions: analysis and reflection, clinical reasons and clinical learning. The total number of items in the scale is 18. The responses to be given for each item are scored as strongly disagree, disagree, not sure, agree, strongly agree. Although there is no cut-off value for the scale, it is interpreted that as the score increases, the level of satisfaction increases. After the simulation evaluation process is completed, students will fill out the scale once based on their self-reports.

SECONDARY OUTCOMES:
Recommendation score | Within 3 weeks after stoma care skill teaching
  The ostomy model developed for this study was created for recommendation scores regarding its use in simulation training. A scoring system will be used to evaluate students' stoma care skill teaching with a wearable ostomy model from 0 to 10. As the student's score increases, it will be interpreted that the model's usability in teaching stoma care skills is high.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Arslan, PhD, Principal Investigator — Director; Havva Yönem Amaç, PhD, Study Chair — Researcher; Sultan Özkan, PhD, Study Chair — Researcher
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.